CLINICAL TRIAL: NCT00520845
Title: A Phase II Trial of Celecoxib Plus Chemotherapy [Docetaxel or Pemetrexed] in Patients With Previously Treated, "COX Dependent" Recurrent Non-Small Cell Lung Cancer
Brief Title: Celecoxib and Docetaxel or Pemetrexed in Treating Patients With Advanced Recurrent Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Leora Horn, MD, Assistant Professor of Medicine; Assistant Director, Educator Development Program; Clinical Director, Thoracic Oncology Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC THO 0730; P30CA068485 (NIH); VU-VICC-THO-0730; VU-VICC-IRB-070723
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib; Docetaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Either docetaxel or pemetrexed given with celecoxib
  Interventions: Drug: celecoxib; Drug: Docetaxel; Drug: pemetrexed disodium; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: celecoxib — 600 mg will be taken by mouth twice a day for 6 weeks then 400 mg twice a day for up to a year after chemotherapy is discontinued in the absence of progression.
Drug: Docetaxel — 75mg/m2 given through a vein over 90 minutes on day 1 of a 3-week cycle
Drug: pemetrexed disodium — 500 mg/m2 through a vein over 90 minutes on day 1 of a 3 week cycle.
Other: laboratory biomarker analysis — Blood collection

SUMMARY:
RATIONALE: Celecoxib may stop the growth of tumor cells by blocking some of the enzymes need for cell growth. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving celecoxib together with docetaxel or pemetrexed may kill more tumor cells.

PURPOSE: This phase II trial is studying how well celecoxib given together with docetaxel or pemetrexed works in treating patients with advanced or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy of celecoxib when administered with standard chemotherapy comprising docetaxel or pemetrexed disodium in patients with advanced, recurrent non-small cell lung cancer (NSCLC) exhibiting cyclooxygenase (COX) dependence.

Secondary

* To determine the overall response rate and time to progression in patients with COX-dependent recurrent NSCLC treated with celecoxib and docetaxel or pemetrexed disodium.
* To determine the effect of celecoxib on the urinary metabolites of PGE_2 , PGI_2, and thromboxane in patients with COX-dependent recurrent NSCLC.
* To correlate changes in urinary PGE-M and survival with intratumoral expression of COX-2, mPGES, and 15-PGDH as assessed by IHC.

OUTLINE: Patients with no prior taxane exposure receive docetaxel IV over 1 hour on day 1; patients with prior taxane exposure or for whom docetaxel treatment is contraindicated receive pemetrexed disodium IV over 10 minutes on day 1. Treatment with docetaxel or pemetrexed disodium repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. All patients receive oral celecoxib twice daily beginning 5-7 days prior to the first docetaxel or pemetrexed disodium infusion and continuing for up to 1 year in the absence of disease progression or unacceptable toxicity.

Patients undergo blood and urine sample collection at baseline and periodically during study for biomarker correlative studies. Urine samples are assessed for PGE-M levels. Blood samples are analyzed for serum celecoxib levels, VEGF, endostatin, and cytokine assays.

After completing the last dose of celecoxib, patients are followed at 4-6 weeks and then every 3 months thereafter for up to 2 years from study entry.

ELIGIBILITY:
Eligibility Criteria:

* Cytologically or histologically confirmed "COX dependent" non-small cell lung cancer.
* COX dependency is defined by change in urinary PGE-M levels following a "run-in" phase of celecoxib.
* Previous treatment with ≤2 different chemotherapy regimens one of which must have been platinum-based (cisplatin or carboplatin) chemotherapy.
* Age ≥18 years
* ECOG PS 0, 1 or 2.
* Measurable or evaluable disease.
* At least 3 weeks post major surgery, chemotherapy or radiotherapy & recovered from all toxicities.
* Expected survival of at least 2 months.
* CNS metastases permitted provided the patient has adequately recovered from radiotherapy includes stereotactic therapy) or surgery.
* Adequate renal function: serum creatinine ≤1.8 mg/dl &/or CrCl >50 cc/min

Eligibility According to Liver Function:

AST:

</= 1.5 ULN-Docetaxel; </= 2.5 ULN-Pemetrexed (Liver parameters to be used for pemetrexed in the absence of proven or radiographically suspected liver metastases.); </= 5.0 ULN-Pemetrexed (Liver parameters to be used for pemetrexed only in the presence of proven or radiographically suspected liver metastases.)

Alk Phosphatase:

</= 2.5 ULN-Docetaxel; </= 2.5 ULN-Pemetrexed (Liver parameters to be used for pemetrexed in the absence of proven or radiographically suspected liver metastases.); </= 5.0 ULN-Pemetrexed (Liver parameters to be used for pemetrexed only in the presence of proven or radiographically suspected liver metastases.)

Total Bilirubin:

</= 1.5 ULN-Docetaxel; </= 1.5 ULN-Pemetrexed (Liver parameters to be used for pemetrexed in the absence of proven or radiographically suspected liver metastases.); </= 2.5 ULN-Pemetrexed (Liver parameters to be used for pemetrexed only in the presence of proven or radiographically suspected liver metastases.)

* Adequate hematologic function: ANC≥1500/mm3 & platelets ≥100,000/mm3
* Female patients cannot be pregnant and must use contraception if of childbearing age
* Lactating women are excluded.
* Peripheral neuropathy must be CTC grade ≤2
* Patients must not currently be on non-steroidal anti-inflammatory agents or other COX-2 inhibitors (Must be off for at least ≤7 days)
* Written informed consent.

Exclusion Criteria:

* More than two prior chemotherapy regimens for recurrent or relapsed NSCLC.
* COX Independent as defined by change in urinary PGE-M levels following a "run-in" phase of celecoxib.
* Previous treatment with both docetaxel and pemetrexed
* History of greater than grade 2 allergic reaction to celecoxib or any other non-steroid anti-inflammatory agent including aspirin, ibuprofen, or indomethacin.
* History of allergy to compounds containing boron or mannitol.
* History of allergy to sulfonamides.
* Concomitant use of Warfarin, but low dose Coumadin allowed for port prophylaxis
* Recent (past 4 weeks) coronary artery bypass graft (CABG) surgery.
* Inadequate organ function:
* Serum creatinine ≥1.8 mg/dl or a calculated CrCl <45 cc/min.
* AST >1.5 upper limits of normal (ULN); alkaline phosphatase >2.5 ULN; & bilirubin >1.5 ULN
* ANC<1500/mm3 & platelets <100,000/mm3
* Active pregnancy or inability or unwillingness to employ appropriate contraception.
* Small cell carcinoma histology.
* Prior malignancy within 5 years of diagnosis of NSCLC. Exceptions include basal cell or non-metastatic squamous cell carcinomas of the skin, cervical carcinoma in situ or FIGO stage I cervical carcinoma, or other cancer history considered not clinically significant by the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-10; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horn, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clnical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened October 2007 and ran to December 2013. All patients were recruited from Vanderbilt-Ingram Cancer Center.
Pre-assignment Details: This study included a "run-in phase" of celecoxib 600 mg BID x 5-7 day, following patient enrollment. Patients with ≥70% decrease in PGE-M level, were considered "COX dependent" and protocol eligible making them eligible for protocol treatment. Patients with <70% decrease in PGE-M level were not eligible.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 23
Completed | 1
Not Completed | 22
Not completed — Death | 3
Not completed — Adverse Event | 4
Not completed — Disease Progression, relapse | 13
Not completed — Withdrawal by Subject | 1
Not completed — Alternative Therapy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 23
Age, Continuous [Mean (Full Range); unit: years] | 63.26 [41 to 79]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Median Survival
Description: Estimated probable duration of life from on-study date to date of death from any cause, using the Kaplan-Meier method with censoring (see analysis population description for additional details)
Time Frame: 2 years from date of registration
Population: All patients are included in the analysis on intention-to-treat basis. Analysis is by Kaplan-Meier method, where death is an event, with censoring for non-expired patients at greater of off-study date or last known alive date.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment Arm
Number analyzed (Participants) | 23
days | 184 [129 to 208]

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate is measured by complete response + partial response. Number of patients in each response category, per RECIST v1.1, summarized as follows for target lesion criteria (see RECIST v1.1 for additional details): complete response (CR),disappearance of target lesions; partial response (PR), >=30% decrease in sum of longest diameter of target lesions; progressive disease (PD), >=20% increase in sum of LD of target lesions or appearance of new lesions; stable disease (SD), insufficient change in target lesions or new lesions to qualify as either PD or SD. Patients are categorized according to the best response achieved prior to occurrence of progressive disease, where best response hierarchy is CR>PR>SD>PD.
Time Frame: On-treatment date to date of disease progression (assessed at 6 weeks up to 2 years)
Population: All patients with best overall response data; patients are excluded if best overall response data is missing or if the patient is not evaluable for best overall response.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 19
participants | 0 [0 to 0.176]

3. Secondary Outcome: Time to Progression
Description: Estimated probable duration from on-study date to date of disease progression, using the Kaplan-Meier method with censoring (see analysis population description for additional details). Disease progression is defined under RECIST v1.1 as >=20% increase in sum of longest diameters of target lesions, unequivocal progression of non-target lesions, or appearance of new lesions.
Time Frame: 2 years from date of registration
Population: All patients are included in the analysis on intention-to-treat basis. Analysis is by Kaplan-Meier method, where progression is an event, with censoring for non-progressed patients at greater of off-study date, last known alive date, or date of death not attributable to disease progression.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment Arm
Number analyzed (Participants) | 23
days | 89 [42 to 386]

4. Other Pre Specified Outcome: Effect of Celecoxib on Urinary Metabolites of PGE2, PG12 and Thromboxane
Time Frame: At 1 year
Population: data is not available. no analysis done
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Changes in Urinary PGE-M and Survival as Assessed by Immunohistochemistry
Time Frame: At 1 year
Population: data is not available. no analysis done
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 17/23
Other Adverse Events (participants affected / at risk) | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=23)
pneumonia, normal ANC (Infections and infestations) | 3 (5)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain abdomen (Gastrointestinal disorders) | 1 (1)
pain pleura (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hemorrhage, lower GI (Gastrointestinal disorders) | 1 (1)
Obstruction - small bowel (Gastrointestinal disorders) | 1 (1)
allergy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
confusion (Psychiatric disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Fever (in the absence of neutropenia) (General disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
Perforation (Gastrointestinal disorders) | 1 (1)
syncope (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 1 (1)
double vision (Eye disorders) | 1 (1)
hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
death (General disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=23)
hyperglycemia (Metabolism and nutrition disorders) | 11 (21)
hyponatremia (Metabolism and nutrition disorders) | 4 (7)
hypoalbuminemia (Metabolism and nutrition disorders) | 3 (5)
ALG, SGPT (Metabolism and nutrition disorders) | 2 (2)
AST, SGOT (Metabolism and nutrition disorders) | 2 (3)
hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
hemoglobinuria (Metabolism and nutrition disorders) | 2 (2)
hemoglobin (Blood and lymphatic system disorders) | 13 (22)
nausea (Gastrointestinal disorders) | 5 (6)
vomiting (Gastrointestinal disorders) | 5 (5)
constipation (Gastrointestinal disorders) | 3 (3)
dyspepsia (Gastrointestinal disorders) | 3 (3)
anorexia (Gastrointestinal disorders) | 2 (2)
gastrointestinal other (Gastrointestinal disorders) | 2 (4)
dysgeusia (taste alteration) (Gastrointestinal disorders) | 2 (2)
pain - thorax (General disorders) | 3 (3)
pain - headache (Nervous system disorders) | 3 (3)
pain - back (Musculoskeletal and connective tissue disorders) | 2 (2)
pain - joint (Musculoskeletal and connective tissue disorders) | 2 (4)
pain - NOS (General disorders) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
pulmonary upper (Respiratory, thoracic and mediastinal disorders) | 2 (2)
dysarthria (Respiratory, thoracic and mediastinal disorders) | 2 (2)
fatigue (General disorders) | 7 (15)
dizziness (Nervous system disorders) | 5 (6)
pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
edema - head and neck (Blood and lymphatic system disorders) | 2 (2)
edema - limb (Blood and lymphatic system disorders) | 2 (2)
fibrillation (Cardiac disorders) | 2 (3)
thrombosis (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes